CLINICAL TRIAL: NCT01693510
Title: Be Healthy in Pregnancy (B-HIP): A Randomized Clinical Trial (RCT) to Study Nutrition and Exercise Approaches for Healthy Pregnancy
Brief Title: Be Healthy in Pregnancy (B-HIP): A Trial to Study Nutrition and Exercise Approaches for Healthy Pregnancy
Acronym: BHIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Dairy Farmers of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BHIP-DFC
Record Dates: First submitted 2012-09-20; First posted 2012-09-26 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2019-03

CONDITIONS: Excessive Weight Gain in Pregnancy as Antepartum Condition; Obesity; Weight Gain; Type 2 Diabetes
Keywords: Excess gestational weight gain (GWG); Obesity; Type 2 diabetes; Elevated fats in the blood; High blood pressure
MeSH Terms: conditions — Obesity; Weight Gain; Diabetes Mellitus, Type 2; Hypertension | interventions — Exercise; Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise and Nutrition Intervention (Experimental): Nutrition intervention: The proposed nutrition plan is a high protein (25% energy) diet providing low fat dairy foods and individualized to energy needs. Dairy foods are accepted by women during pregnancy as a healthy choice (from pilot study) and in our recent birth cohort study, women consumed an average of 3 or more servings of dairy per day. Exercise intervention: Most previous studies and published guidance focus on aerobic exercise such as walking as it is the easiest physical activity to implement in pregnancy in terms of setting goals of steps and monitoring of adherence using accelerometer-type devices. Walking is also the most practical since women reduced moderate and vigorous physical activity during pregnancy but levels of walking were maintained.
  Interventions: Behavioral: Exercise and Nutrition Intervention
- Usual Prenatal Care (No Intervention): Mothers in the Control Group will be followed by their primary care provider and have usual access to public health. In addition, women will have the opportunity to attend one focus group session exploring women's experiences with nutrition, exercise, and weight gain in pregnancy.

INTERVENTIONS:
Behavioral: Exercise and Nutrition Intervention — Both Intervention and Control participants and their care providers receive the new Health Canada guide on Healthy Weight Gain During Pregnancy. For the Experimental Group, the exercise intervention includes a custom-designed pregnancy-specific group walking class of 30-60 min. 1x/week and a prescribed at-home walking program to reach 10,000 steps/day. The nutrition intervention is a high protein (25% energy) low-fat dairy food plan designed to meet energy needs and with individualized counselling.
  Arms: Exercise and Nutrition Intervention

SUMMARY:
Weight gained during pregnancy is referred to as gestational weight gain (GWG). Excess GWG is a widespread problem that occurs in 55-75% of Canadian women who enter pregnancy overweight or obese (a group that represents over 50 % of all pregnant women) and about 40% women of normal weight. Excess GWG is associated with complications of pregnancy, such as post-partum weight retention, type 2 diabetes, elevated fats in the blood, and high blood pressure and may also lead to problems with the health of the newborn child. Our research aims to find ways to control GWG by developing new and practical approaches to diet and exercise targeted to overweight pregnant women that hold promise of improving their health both during pregnancy and thereafter. The experimental intervention is a diet of higher protein provided by dairy foods combined with an exercise program modified to the abilities of overweight pregnant women; and the control is the usual advice given by their primary care providers, information on healthy pregnancy from Health Canada, and a focus group session exploring women's experiences with exercise, nutrition, and gestational weight gain. The results of this study will allow us to design future large clinical studies in all pregnant women to help control the weight gain in all pregnant women.

DETAILED DESCRIPTION:
This will be a 2-arm randomized 1-site trial. Recruitment will be within the community care clinics by poster and flyer advertisements.

Primary research question: Among pregnant women, does introducing a structured and monitored nutrition and exercise program (treatment) in early pregnancy compared with Usual Prenatal Care (control) increase the likelihood of attaining gestational weight gain within the Institute of Medicine (IOM) guidelines over the pregnancy period?

Experimental and Control groups: Both groups of mothers and their health care providers will be given the Health Canada materials on "Healthy Weight Gain during Pregnancy", "Eating Well with Canada's Food Guide" and the "Pregnancy Weight Gain Calculator". Baseline information will be recorded for eligible and consenting women after which they will be randomized to Experimental or Control group. Nutrition intake, physical measures and physical activity will be recorded at baseline, 26-28 weeks and 36-38 weeks of gestation and 6 months post partum in the same manner for both groups. All mothers will receive the study promotional materials and small incentives. Also, all mothers will be followed by their primary care provider and have usual access to Public Health.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant females > 18 years of age with singleton pregnancies (either nulliparous or multiparous); less than 20 weeks gestation; pre-pregnancy BMI of >25 and < 40 kg/m2 (owing to the fact that severe obesity with BMI> 40 may have limitations with respect to physical activity); plans to deliver at a Hamilton Health Sciences, St. Joseph's Healthcare Hamilton, Joseph Brant Hospital or by home birth but willing to attend research visits at the McMaster University Medical Centre site; approval of primary care provider; and able to provide signed informed consent.

Exclusion Criteria:

* Unable to understand some English; currently breastfeeding previous child; pregnancy resulting from in vitro fertilization; known contraindications to exercise as recommended by the Canadian clinical practice guidelines for pregnancy; severe chronic gastrointestinal diseases or conditions; refusal to consume dairy foods due to intolerance or dislike; any significant heart, kidney, liver or pancreatic diseases; pre-existing diabetes; or a depression score above 13 on the validated Edinburgh Depression scale as that is indicative of severe depression and should be referred for treatment; currently smoking.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2012-11-12 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Gestational weight gain within IOM guidelines | Change from baseline at 38 weeks gestation
  Among pregnant women (population), does introducing a structured and monitored nutrition and exercise program (treatment) in early pregnancy compared with Usual Prenatal Care (control) increase the likelihood of attaining GWG within the IOM guidelines (outcome) over the pregnancy period?

SECONDARY OUTCOMES:
Bone outcomes | 6 months post-partum
  Bone status in mothers and infants at 6 months after delivery will be assessed against reference data for bone mineral content (infants) or bone mineral density (mothers) and anthropomorphic outcomes in babies (weight and height).

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A. Atkinson, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University Medical Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palacios C, Kostiuk LL, Cuthbert A, Weeks J. Vitamin D supplementation for women during pregnancy. Cochrane Database Syst Rev. 2024 Jul 30;7(7):CD008873. doi: 10.1002/14651858.CD008873.pub5. PMID 39077939
- [Derived] Maran A, Atkinson SA, Bertram V, Vanniyasingam T, Thabane L, Mottola MF, Phillips SM; BHIP study team. Exploring comparative assessment of adiposity measures during pregnancy and postpartum. Clin Nutr ESPEN. 2022 Jun;49:365-371. doi: 10.1016/j.clnesp.2022.03.021. Epub 2022 Mar 23. PMID 35623838
- [Derived] Perreault M, Atkinson SA, Meyre D, Fusch G, Mottola MF; BHIP Study Team. Summer Season and Recommended Vitamin D Intake Support Adequate Vitamin D Status throughout Pregnancy in Healthy Canadian Women and Their Newborns. J Nutr. 2020 Apr 1;150(4):739-746. doi: 10.1093/jn/nxz276. PMID 31732740